CLINICAL TRIAL: NCT04279522
Title: The MOOD Study - External Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) for the Treatment of Major Depressive Disorder (MDD)
Acronym: MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-201-MOOD
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: MDD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group 1 - active stimulation (Experimental)
  Interventions: Device: Relivion®DP- Active
- Group 2 - sham stimulation (Placebo Comparator)
  Interventions: Device: Relivion®DP- Sham

INTERVENTIONS:
Device: Relivion®DP- Active — Relivion®DP- Active stimulation device
  Arms: Group 1 - active stimulation
Device: Relivion®DP- Sham — Relivion®DP- Sham stimulation device
  Arms: Group 2 - sham stimulation

SUMMARY:
The MOOD study will evaluate the safety and efficacy of a noninvasive, self-administered external Combined Occipital and Trigeminal Neurostimulation (eCOT-NS) treatment for Major Depressive Disorder (Relivion®DP).

This is a prospective, multi-center, 2-arm randomized, double-blind, parallel-group, sham-controlled study.

The study will include the following stages:

1. Screening, Eligibility evaluation and Randomization to Relivion®DP vs. Sham control (1:1 randomization) (Baseline - Day 0).
2. Daily treatment period: Active/Sham (Group A/B) treatment protocol (Baseline to end of 8 weeks).
3. Open label phase: Active treatment period of additional 8 weeks.

After completion of the open label period the subject's participation in the study will be over.

DETAILED DESCRIPTION:
The study will include the following study visits & phases:

* Visit 1- Screening (Day (-14)-0) - Screening & Preliminary Eligibility Assessment.
* Visit 2- Baseline (Day (-4)-0) - Eligibility, baseline assessment, Randomization to Relivion®DP vs. Sham control (1:1 randomization) and training.
* Double blind phase (Day 0 to day 56±7)- 5-7 days a week treatment: Active/Sham (Group A/B) treatment protocol.
* Visit 3- Follow Up Visit (day 28±7)- MDD assessment.
* Visit 4- End of Double-Blind phase (day 56±7)- MDD assessment.
* Open label phase- Active treatment period: According to HDRS response in DB phase, in between Maintenance treatment 3-4 times a week and up to 5-7 days a week of intensified treatment (Day 56±7 to day 112±7)
* Visit 5- follow up visit (day 84±7) - MDD assessment.
* Visit 6- End of study (day 112±7)- MDD assessment and end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-70 years of age:

   1. Up to 124 randomized subjects aged 22-70
   2. Up to 36 randomized subjects aged 18-21
2. Primary diagnosis of unipolar major depressive disorder by DSM-V criteria.
3. Current MDD episode lasts up to three years.
4. Score on the Hamilton Depression Rating Scale (HDRS21) ≥ 20
5. Symptoms of current major depressive episode that, as determined by the Investigator, for the current episode and according to the Antidepressant Treatment Resistance Form (ATRF) or Antidepressant Treatment Intolerance Form (ATIF):

   * Did not respond or have insufficiently responded by less than 50% improvement; dose and duration defined & rated at minimum confidence level 3 on the ATRF;
   * Did not respond or has insufficiently responded to at least one but no more than four adequate trials of antidepressant medications (4 ≥ ATRF ≥1) or
   * Did not respond or has insufficiently responded due to poor tolerability to at least two inadequate antidepressant medication trials (ATIF ≥2).
6. Subject must be on at least one (1) antidepressant medication (minimum therapeutic dose not required if tolerability precluded further dose titration) and is willing to remain on the same daily dose of antidepressant medication(s) for a minimum of 28 days prior to randomization and thereafter for the duration of the study.
7. For subjects receiving current depression focused psychotherapy: psychotherapy initiated at least 1 month prior to baseline visit with a stable frequency of visits regimen, in the opinion of the Investigator.
8. Subject is able to provide written Informed Consent and is capable of complying with the specified study requirements, as determined by the Investigator.
9. Subject has cognitive and/or motor skills needed to operate a smartphone and can be contacted by phone, as determined by the Investigator.

Exclusion Criteria:

1. History of intracranial surgery.
2. Current denervation in one or more of the following: the supraorbital or supratrochlear branches of the trigeminal nerve, or the greater occipital branch of the occipital nerve.
3. An implanted neurostimulators or any implanted metallic or electronic device in the head, a cardiac pacemaker or an implanted or wearable defibrillator, except for dental implants.
4. Skin lesion, scars, or inflammation at the region of the stimulating electrodes.
5. Subjects with a history of traumatic brain injury (TBI), defined as a disruption in the normal function of the brain that can be caused by a bump, blow, or jolt to the head, or penetrating head injury, within 3 months of study enrollment.
6. Pregnancy or Lactation.
7. Women of reproductive age not using a reliable contraceptive method as determined by the Investigator.
8. In the opinion of the Investigator, subjects with a psychiatric history consistent with, suspicious for, or diagnostic of, bipolar depression or depression associated with psychosis.
9. Borderline personality disorder, defined by DSM-V criteria, that in the judgement of the Investigator is likely to complicate the assessment of clinical response to study treatments or limits the patient's ability to comply with study procedures
10. Subjects who, within one (1) year of study enrollment, have a history consistent with, suspicious for or diagnostic of, any of the following: psychosis, psychotic disorder, schizophrenia or schizoaffective disorder, in the opinion of the Investigator.
11. Subjects who demonstrate or have a history of any cognitive disorder or impairment, memory loss, dementia, confusion or delirium that, in the opinion of the Investigator, may compromise the integrity of the study data or impact the ability of the subject to comply with the study requirements.
12. Past 12 months active suicidal intent or plan as defined by a "yes" answer to Q4 or Q5 on the Columbia-Suicide Severity Rating Scale, (C-SSRS) or with a history of suicide attempt in the past twelve months.
13. Subjects currently (past month) meeting diagnostic criteria for Obsessive-Compulsive Disorder or post-traumatic stress disorder and that is their primary diagnosis.
14. Subjects meeting the DSM-V criteria for alcohol use disorder or other substance use disorder (not including tobacco/nicotine) within six (6) months prior to study enrollment.
15. The subject has any past or present medical condition, disease, illness, disorder or injury that, in the opinion of the Investigator, may reduce or hinder the subject's ability to fully comply with all study requirements for the duration of the study or may confound the integrity of the study data.
16. Participation in a previous study with the Relivion®DP or the Relivion® device.
17. Treatment with Transcranial Magnetic Stimulation (TMS) in the past 6 months.
18. Current treatment with any other approved or investigational brain stimulation therapies (i.e. Vagus or trigeminal nerve Stimulation, tDCS, TES).
19. Failure to receive clinical benefit from an adequate trial of ECT in the current or a past depressive episode in the opinion of the Investigator.
20. Subject having received Botox treatment in the head or neck region within 90 days prior to study enrollment.
21. Subject having received supraorbital or occipital nerve blocks within 1 month prior to enrollment.
22. Head circumference smaller than 51 centimeters or larger than 60 centimeters.
23. Current neurological condition or disease which, in the opinion of the investigator, is likely to manifest a depressive syndrome or symptoms that would substantially confound the diagnosis or serial assessment of major depressive disorder.
24. Subjects participating in other clinical trials evaluating experimental treatments or procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carpenter, MD, Principal Investigator — Butler Hospital, Brown Department of Psychiatry and Human, RI, USA Behavior,
Locations (13):
- United States (12):
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - UCLA Semel Institute for Neuroscience and Behaviour, Los Angeles, California
  - San Marcus Research Clinic, Miami Lakes, Florida
  - K2 Medical Research Tampa, Tampa, Florida
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Sheppard Prat Health system, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of North Carolina, Department of Psychiatry, Chapel Hill, North Carolina
  - Butler Hospital/Brown University, Providence, Rhode Island
  - VA Providence Healthcare System, Providence, Rhode Island
  - MUSC Institute of Psychiatry, Charleston, South Carolina
  - Brain Health Consultants and TMS Center, Houston, Texas
- Ichilov Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1: Double Blind Phase
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Started (As randomized 62 Active and 62 Sham. As treated, there were 63 Active and 61 Sham since we had one randomization error when a subject received by the site team the wrong device type by mistake.) | 62 | 62
Completed (out of the 104 subjects completing the DB phase, only 96 started the OLE phase. 3 subjects (2 Active, 1 Sham) decided not to participate (OLE phase was optional). 1 subject (Sham) did not participate as the site closed the research center. 4 subjects (3 Active, 1 Sham) did not proceed to the OLE phase due to not reaching DB phase compliance.) | 51 | 53
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Protocol Violation | 1 | 0
Period: Period 2: Open Label Phase
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Started | 46 | 50
Completed | 42 | 43
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (13.14) | 48.1 (13.14) | 48.6 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 89
  Male | 19 | 16 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 44 | 44 | 88
  African or African-American | 2 | 3 | 5
  Asian | 2 | 1 | 3
  American Indian or Alaska Native | 0 | 1 | 1
  other | 14 | 12 | 26
  not reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 121
  Israel | 1 | 2 | 3
Number of antidepressant medications with none or insufficient response in the current episode [Mean (Standard Deviation); unit: Number of antidepressant medications] — antidepressants medication history within the subjects' current major depressive episode that, as determined by the Investigator and according to the Antidepressant Treatment Resistance Form (ATRF), the subjects did not respond to or have insufficiently responded by less than 50% improvement; dose and duration defined and rated at minimum confidence level 3 on the ATRF.
  Number of antidepressant medications | 1.8 (0.97) | 1.8 (0.89) | 1.8 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Depressive Symptoms, Measured by HDRS17 Total Score
Description: Mean change in depressive symptoms, measured by HDRS17 total score, from baseline to week-8 post treatment initiation.
  The HDRS-17 (17-item Hamilton Depression Rating Scale) is a widely used, clinician-administered questionnaire designed to assess the severity of depressive symptoms. Total score ranges from 0 to 52-higher scores indicate more severe depression.
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
units on a scale | -8.62 (0.8476) | -6.01 (0.8257)

2. Secondary Outcome: Percentage of Responder Participants
Description: Proportion of responder subjects- defined as the percent of subjects achieving at least 50% reduction from baseline in their HDRS17 scale 8 weeks post Relivion®DP treatment initiation.
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
Participants | 15 | 9

3. Secondary Outcome: Percentage of Subjects Achieving Remission
Description: Proportion of subjects achieving remission- defined as the percent of subjects with HDRS17 score≤7 at 8 weeks post treatment initiation
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
Participants | 10 | 3

4. Secondary Outcome: Mean Change in Depressive Symptoms, Measured by MADRS Total Score
Description: Mean change in depressive symptoms, measured by MADRS total score, from baseline to week-8 post treatment initiation.
  The MADRS stands for the Montgomery-Åsberg Depression Rating Scale. It is a clinician-administered tool used to assess the severity of depressive symptoms, particularly in clinical trials and psychiatric evaluations. Contains 10 items, each scored from 0 to 6, with a total possible score ranging from 0 to 60. Higher scores indicate more severe depression.
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
units on a scale | -10.18 (1.2874) | -8.09 (1.2611)

5. Other Pre Specified Outcome: Mean Change in Depressive Symptoms Severity and Improvement Scores
Description: Mean Change in the severity and improvement scores - Clinical Global Impression scales (CGI-S and CGI-I) at 8 weeks post treatment initiation.
  he CGI-S (Clinical Global Impression - Severity) and CGI-I (Clinical Global Impression - Improvement) are two components of the CGI scale, a brief, standardized assessment used by clinicians to rate the severity of a patient's illness and their improvement over time, typically in clinical trials and psychiatric practice. both on a Scale of 1 to 7. higher score on the CGI-S indicate more severe depression. Higher score on the CGI-I indicates worsening depression.
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
units on a scale
  CGI-S | -1.15 (0.1703) | -0.85 (0.1661)
  CGI-I | 3.51 (0.2021) | 4.05 (0.1975)

6. Other Pre Specified Outcome: Mean Change in Quick Inventory of Depressive Symptomatology Self-rated Score
Description: Mean Change from baseline in total score of the Quick Inventory of Depressive Symptomatology self-rated (QIDS-SR-16) score at 8 weeks post treatment initiation.
  The QIDS-SR-16 stands for the Quick Inventory of Depressive Symptomatology - Self-Report, 16-item version. It is a self-administered questionnaire designed to assess the severity of depressive symptoms in patients. Total score range: 0 to 27. Higher scores indicate more severe depression.
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
units on a scale | -4.59 (0.6407) | -3.57 (0.6294)

7. Other Pre Specified Outcome: Mean Change in Depressive Symptoms, Measured by HDRS21 Total Score
Description: Mean change in depressive symptoms, measured by HDRS21 total score, from baseline to week-8 post Relivion®DP treatment initiation.
  The HDRS-21, or 21-item Hamilton Depression Rating Scale, is an extended version of the original Hamilton Depression Rating Scale (HDRS17). It is a clinician-administered tool designed to assess the severity of depressive symptoms in patients diagnosed with major depressive disorder (MDD). Total score range: 0 to 64. higher scores indicate more severe depression.
Time Frame: 8 weeks from treatment initiation
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation
Number analyzed (Participants) | 47 | 50
units on a scale | -8.86 (0.8916) | -6.11 (0.8658)

ADVERSE EVENTS:
Time Frame: throughout the study conduct from the point of enrollment, for each enrolled subject up to 18 weeks post treatment initiation. per protocol each of the treatment periods (Double Blind and Open Label) lasted up to 9 weeks.
Description: Safety of the study device following study treatment: incidence of adverse events and serious adverse events related or unrelated to the study device.
Groups:
- Open Label Active Stimulation: Relivion®DP- Active stimulation device
Arm/Group | Group 1 - Active Stimulation | Group 2 - Sham Stimulation | Open Label Active Stimulation
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 1/96
Other Adverse Events (participants affected / at risk) | 18/62 | 20/62 | 29/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Active Stimulation (N=62) | Group 2 - Sham Stimulation (N=62) | Open Label Active Stimulation (N=96)
worsening of depression symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — The participant requested to be hospitalized, and the Investigator decided to follow through with her request. The event occurred during the open-label phase of the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Active Stimulation (N=62) | Group 2 - Sham Stimulation (N=62) | Open Label Active Stimulation (N=96)
Headache (Nervous system disorders) | 5 (19) | 2 (2) | 5 (12)
Redness/ indentation on forehead (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scalp itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation/ erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Stinging sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Worsening depression symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Pressure in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
AEs definitely not related to the study device (General disorders) | 13 (19) | 16 (21) | 22 (26)
Unpleasant sensation during treatment (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall have the right to publish the results and information about the results. PI agree to submit any proposed publication to Sponsor for review and approval at least 60 days prior to submitting to a publisher. Sponsor shall respond in writing within 45 days of its receipt and have the right to require PI to (a) remove Confidential Information; (b) delay the proposed Publication for an additional ninety (90) days to enable Sponsor to seek patent application or other proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT04279522/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT04279522/SAP_001.pdf